CLINICAL TRIAL: NCT01085734
Title: A 6-Month, Single Site, Masked, Randomized,Controlled Study to Assess Efficacy of Osurdex as Adjunct to Avastin Compared With Avastin Alone in the Treatment of Patients With Macular Edema Due to Central or Branch Retinal Vein Occlusion
Brief Title: Single Site, Masked, Randomized, Controlled Study to Assess Efficacy of Osurdex as Adjunct to Avastin Compared With Avastin Alone in the Treatment of Patients With Macular Edema Due to Central or Branch Retinal Vein Occlusion
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Maturi, Raj K., M.D., P.C. (Individual)
Responsible Party: Principal Investigator, Raj K. Maturi, MD, President, Maturi, Raj K., M.D., P.C.
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OA001
Record Dates: First submitted 2010-03-10; First posted 2010-03-12 (Estimated); Results first posted 2014-04-21 (Estimated); Last update posted 2014-04-21 (Estimated); Status verified 2014-03

CONDITIONS: Retinal Vein Occlusions
MeSH Terms: conditions — Retinal Vein Occlusion | interventions — Bevacizumab

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Active Comparator): Group 1 receives Avastin at baseline followed by sham Osurdex at week 1. Additional Avastin based on macular edema
  Interventions: Drug: Avastin
- Group 2 (Active Comparator): Group 2 receives Avastin at baseline followed by Osurdex at week 1. Retreatment with Avastin based on macular edema
  Interventions: Drug: Osurdex; Drug: Avastin

INTERVENTIONS:
Drug: Avastin — 1.25mg intravitreally
  Arms: Group 1
Drug: Osurdex — 0.7mg intravitreally
  Arms: Group 2
Drug: Avastin — 1.25mg intravitreally
  Arms: Group 2

SUMMARY:
Comparative study to see if treating with Osurdex in addition to Avastin in patients with retinal vein occlusions helps increased visual acuity outcomes

ELIGIBILITY:
Inclusion Criteria:

* male or female age 18 years or older
* Branch retinal vein occlusion or central retinal vein occlusion of less than one year duration
* Best correct visual acuity of greater than 24 and less than 80
* Presence of macular edema defined as OCT central subfield thickness of >250

Exclusion Criteria:

* intravitreal anti-VEGF treatment in study eye within six weeks of baseline
* intravitreal steroid treatment in the study eye within eight weeks of baseline visit
* PRP in the study eye within 4 month of baseline visit
* Active iris neovascularization in study eye
* Uncontrolled systemic disease
* Known history of IOP elevation in response to corticosteroid treatment that is not controlled on 2 glaucoma medications

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2010-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raj K Maturi, MD, Principal Investigator — Raj K. Maturi, MD, PC
Locations (1):
- Raj K. Maturi, MD, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at a single center. The first subject for this study was screened on 18MAR2010 and enrolled on 26MAR2010. The subjects were existing patients in our medical clinic.
Pre-assignment Details: In total there were 10 screen failures; 4 did not meet the visual acuity requirements,3 did not meet the OCT requirements. One subject withdrew consent prior to randomization and one withdrew prior to randomization due to health issues
Groups:
- Group 1: Group 1 receives intravitreal Avastin at baseline followed by sham Osurdex at week 1. Additional treatment with Avastin was given at monthly intervals when the OCT central subfield thickness was greater than 250 microns. Retreatment with sham Osurdex occurred at month 4 one week after Avastin treatment if central edema was greater than 250 micros
- Group 2: Group 2 receives intravitreal Avastin at baseline followed by Osurdex at week 1. Retreatment with Avastin was given at monthly intervals wehn the OCT central subfield thickness was greater than 250 microns. Retreatment with Osurdex occurred at month 4 one week after Avastin treatment if central edema was greater than 250 microns.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 15 | 15
Completed | 14 | 11
Not Completed | 1 | 4
Not completed — Adverse Event | 0 | 2
Not completed — Death | 1 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Group 1: Group 1 receives intravitreal Avastin at baseline followed by sham Osurdex at week 1. Additional treatment with Avastin was given at monthly intervals when the OCT central subfield thickness was greater than 250 microns. Retreatment with sham Osurdex occurred at month 4 one week after Avastin treatment if cnetral edema was greater than 250 micros
- Group 2: Group 2 receives intravitreal Avastin at baseline followed by Osurdex at week 1. Retreatment with Avastin was given at monthly intervals wehn the OCT central subfield thickness was greater than 250 microns. Retreatment with Osurdex occurred at month 4 one week after Avastin treatment if cnetral edema was greater than 250 microns.
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 6 | 4 | 10
  >=65 years | 9 | 11 | 20
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (13) | 69 (19) | 68 (16)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 10 | 8 | 18

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline Visual Acuity at 6 Months
Description: Visual Acuity was measured with ETDRS visual acuity test. Unit of measure is based on the ETDRS letter score scale, 0-97, where 0 = worst and 97 = best.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ETDRS score
Groups:
- Group 1: Group 1 receives intravitreal Avastin at baseline followed by sham Osurdex at week 1. Additional treatment with Avastin was given at monthly intervals when the OCT central subfield thickness was greater than 250 microns. Retreatment with sham Osurdex occurred at month 4 one week after Avastin treatment if central edema was greater than 250 microns.
- Group 2: Group 2 receives intravitreal Avastin at baseline followed by Osurdex at week 1. Retreatment with Avastin was given at monthly intervals when the OCT central subfield thickness was greater than 250 microns. Retreatment with Osurdex occurred at month 4 one week after Avastin treatment if central edema was greater than 250 microns.
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 11
ETDRS score | 2.3 (7.7) | 0.1 (13.3)

2. Secondary Outcome: Number of Injections Needed
Description: number of Avastin and Ozurdex injections needed
Time Frame: baseline to 6 months
Measure: Number; unit: injections
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 11
injections | 14 | 11

3. Secondary Outcome: Change in Macular Thickness and Macular Volume
Description: OCT central subfield thickness measured in microns
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: microns
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 14 | 11
microns | 45.4 (100.1) | -55.6 (39.7)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Group 1 | Group 2
Serious Adverse Events (participants affected / at risk) | 4/15 | 3/15
Other Adverse Events (participants affected / at risk) | 13/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=15) | Group 2 (N=15)
breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
esophageal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
viral influenza (Immune system disorders) | 0 (0) | 1 (1)
osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
organ transplant rejection (Immune system disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=15) | Group 2 (N=15)
worsening of cataract (Eye disorders) | 1 (1) | 3 (3)
worsening of hypertension (Cardiac disorders) | 1 (1) | 1 (1)
back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 1 (1) | 0 (0)
osteoporosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
generalized weakness (General disorders) | 0 (0) | 1 (1)
increased intraocular pressure (Eye disorders) | 1 (1) | 1 (1)
worsening of epiretinal membrane (Eye disorders) | 0 (0) | 1 (1)
subconjunctival hemorrhage (Eye disorders) | 1 (1) | 0 (0)
urinary incontinence (Renal and urinary disorders) | 0 (0) | 1 (1)
contusion left foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
sinusitis (Ear and labyrinth disorders) | 1 (1) | 0 (0)
inner ear infection (Ear and labyrinth disorders) | 0 (0) | 1 (1)
vitreous floaters (Eye disorders) | 0 (0) | 2 (2)
infection left foot (Infections and infestations) | 0 (0) | 1 (1)
auditory disturbance (Ear and labyrinth disorders) | 0 (0) | 1 (1)
puncture wounds to hands (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
blurry vision (Eye disorders) | 0 (0) | 1 (1)
tooth infection (Infections and infestations) | 1 (1) | 0 (0)
discomfort right eye (Eye disorders) | 1 (1) | 0 (0)
nonfunctioning gallbladder (Hepatobiliary disorders) | 0 (0) | 1 (1)
anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
cholescystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
knee pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
headache (General disorders) | 0 (0) | 1 (1)
nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No